CLINICAL TRIAL: NCT07361341
Title: Culturally Tailored Program for Food-Insecure Adults With Type 2 Diabetes: The SPICE-D Study (Support for People Through Inclusive Cultural Eating for Diabetes)
Brief Title: Culturally Tailored Program for Food-Insecure Adults: SPICE-D
Acronym: SPICE-D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00141289
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus (T2D)
Keywords: type 2 diabetes mellitus; culture; nutrition; Spanish; food insecurity
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Food Bundles (Experimental): active patients of the Community Care Clinic with diagnosis of Type 2 diabetes or pre-diabetes with an hemoglobin A1c of >/= 9.5% who are food insecure
  Interventions: Other: Food Bundle Intervention

INTERVENTIONS:
Other: Food Bundle Intervention — Culturally tailored food bundles containing Hispanic-friendly ingredients that support diabetes management, as well as recipe resources and cooking guides designed for various literacy levels.

SUMMARY:
The goal of this pilot intervention study is to learn if culturally appropriate food bundles and nutrition education can help people with diabetes who struggle to afford healthy food in patients with diabetes receiving care at Community Care Clinic in Winston-Salem, NC. The main questions we hope to answer are:

1. Can providing culturally appropriate foods and recipes improve how people cook and prepare meals at home?
2. Can this approach improve people's nutrition knowledge and help them better manage their diabetes?
3. Can this approach improve overall health outcomes for people with diabetes who face food insecurity?

Participants will:

1. Complete an initial interview and survey about their food security, health challenges, and social needs
2. Receive culturally appropriate food bundles designed for their community
3. Receive easy-to-use educational materials including recipes and cooking guides that match their reading level
4. Complete follow-up surveys at 3 months and 6 months to track any changes in their cooking habits, nutrition knowledge, diabetes management, and health

DETAILED DESCRIPTION:
The purpose of this hybrid study is to examine the relationship between food insecurity and health outcomes among predominantly Hispanic, low-income patients at the Community Care Clinic (CCC), and to evaluate the impact of culturally tailored food interventions on diabetes management and overall health. Using retrospective chart review and prospective cohort analysis, this research will assess how food insecurity affects key health indicators including glycemic control (HbA1c), blood pressure, body mass index, and healthcare utilization patterns. Qualitative interviews also will elucidate patient perspectives of their care, their food choices, and their experiences managing diabetes. Through the provision of culturally familiar food bundles and recipe resources over a three-month period, this study aims to identify effective, community-centered nutritional strategies that address both the structural barriers and cultural dimensions of food insecurity in this vulnerable population. The findings will inform evidence-based interventions to improve diabetes care and reduce health disparities among uninsured, low-income patients at the CCC and similar safety-net clinics serving marginalized communities.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years at the time of the first clinic visit during the study period; regardless of sex, gender, race, or ethnicity
* Active patients of the Community Care Clinic (CCC) who received at least one clinical encounter between January 1, 2024 and December 31, 2024; with at least one scheduled follow-up appointment during the prospective study period
* Meet CCC's standard eligibility criteria: Uninsured status (no health insurance coverage); Family income ≤250% of the Federal Poverty Level; Resident of Forsyth County, North Carolina, or surrounding service area
* Completed at least one validated food insecurity screening tool during the study period as part of routine clinical care
* Medical record contains at least one documented measurement for any of the primary outcome variables (body mass index, blood pressure, HbA1c, or healthcare utilization metric)
* Documented diagnosis of Type 2 diabetes (ICD-10: E11.x) OR; Pre-diabetes diagnosis (ICD-10: R73.03) with a hemoglobin A1c ≥9.5%
* Reside within designated pickup/delivery zones for food bundle distribution (primary zip codes: 27101, 27105, 27107, and adjacent service areas)
* Able and willing to provide written informed consent (available in English and Spanish)
* Able to participate in baseline and follow-up assessments either in English or Spanish (the two primary languages at CCC)

Exclusion Criteria:

* Unable to speak proficiently in English or Spanish, as this study and the CCC staff are equipped only to provide services in English and Spanish languages.
* Have known food allergies (documented in the electronic medical record and/or self-reported to CCC or study staff) that may preclude participation in the food bundle program inherent to this protocol.
* Have incomplete records. Medical charts with missing or incomplete demographic information (age, gender) that cannot be verified through other sources
* Patients who were pregnant at any point during the study period (due to expected physiological changes in weight, blood pressure, and glucose metabolism that would confound outcome measurements)
* Patients with documented terminal illness or hospice care during the study period, as their health trajectory and care priorities differ fundamentally from the general population
* Transient patients. Patients who received only one-time urgent/emergent care without established continuity of care at CCC (defined as <2 visits during study period)
* Type 1 diabetes (ICD-10: E10.x) - requires different dietary management; End-stage renal disease requiring dialysis (special dietary restrictions); Active eating disorder diagnosis; Severe food allergies that would limit ability to safely consume food bundle contents; Recent bariatric surgery (<12 months)
* Documented cognitive impairment or intellectual disability that would impair ability to provide informed consent or participate meaningfully in intervention without caregiver support
* Currently enrolled in other intensive nutrition intervention studies or food prescription programs that would confound assessment of the intervention's independent effects
* Primary language other than English or Spanish
* Plans to move outside of CCC's service area or discontinue care at CCC within the 6-month study period
* Physical disabilities, literacy barriers, or other factors that would prevent completion of baseline or follow-up survey instruments, unless accommodations can be reasonably made

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | Baseline
  HbA1c levels will be obtained via the medical record to indicate glycemic control in patients with diabetes.
Hemoglobin A1c | Month 3
  HbA1c levels will be obtained via the medical record to indicate glycemic control in patients with diabetes.
Hemoglobin A1c | Month 6
  HbA1c levels will be obtained via the medical record to indicate glycemic control in patients with diabetes.
Self-efficacy in diabetes management | Baseline
  Self-efficacy in diabetes management will be assessed using questions adapted from the Self Efficacy for Managing Diabetes Scale. The instrument includes 8 questions assessing how secure patients feel in managing their diabetes. Questions include a Likert scale ranging from 1 to 10, where 1 represents low self efficacy and 10 represents high self efficacy.
Self-efficacy in diabetes management | Month 3
  Self-efficacy in diabetes management will be assessed using questions adapted from the Self Efficacy for Managing Diabetes Scale. The instrument includes 8 questions assessing how secure patients feel in managing their diabetes. Questions include a Likert scale ranging from 1 to 10, where 1 represents low self efficacy and 10 represents high self efficacy.
Self-efficacy in diabetes management | Month 6
  Self-efficacy in diabetes management will be assessed using questions adapted from the Self Efficacy for Managing Diabetes Scale. The instrument includes 8 questions assessing how secure patients feel in managing their diabetes. Questions include a Likert scale ranging from 1 to 10, where 1 represents low self efficacy and 10 represents high self efficacy.

SECONDARY OUTCOMES:
Body Mass Index | Baseline, 3 months, 6 months
  Body Mass Index will be assessed from height and weight data in the electronic medical record.
Patient perceptions of intervention | Baseline, 3 months, 6 months
  Qualitative interviews will assess participant perceptions of the intervention, the food received, and thoughts about diabetes management. Each interview will include 20 questions. Information from the interviews will be qualitatively coded to develop themes reflecting participants' collective perceptions.
Diabetes literacy | Baseline, 3 months, 6 months
  Diabetes literacy will be assessed via a series of questions adapted from the Diabetes Literacy Scale to gauge participants' knowledge of standard type 2 diabetes information and diabetes related nutrition. The questionnaire includes 15 items scored on a 5 point Likert scale where 1 reflects low literacy and 5 reflects high literacy.
Number of Emergency Department Visits | baseline, 3 months, 6 months
  Data from the electronic medical record will be used to calculate the number of emergency department visits attended for each participant during the previous 3 months. Data will be total numeric counts of emergency department visits.
Number of Missed Appointments | baseline, 3 months, 6 months
  Data from the electronic medical record will be obtained to provide the number of missed medical appointments at the Community Care Clinic for each patient during the previous 3 months. Data will be numeric counts of the total number of missed visits.
Diastolic and Systolic Blood Pressure (mm/Hg) | baseline, 3 months, 6 months
  Diastolic and Systolic blood pressure (mm/Hg) will be obtained from the electronic medical record for each patient corresponding to the date of their routine medical visit at the Community care Clinic.

OTHER OUTCOMES:
Difference in hemoglobin A1c levels between food-secure and food-insecure groups | up to 12 months
  Retrospective chart review will be used to determine the difference in hemoglobin A1c of patients who are food-secure and food-insecure.

CONTACTS AND LOCATIONS:
Overall Officials: Megan B Irby, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No